CLINICAL TRIAL: NCT02723422
Title: Intensive Versus Usual Home-based Physical Therapy to Promote Functional Recovery After Transcatheter Aortic Valve Replacement (TAVR): A Pilot Randomized Trial
Brief Title: Transcatheter Aortic Valve Replacement (TAVR)-Pilot Trial
Acronym: TAVR-PT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-01098
Record Dates: First submitted 2016-03-09; First posted 2016-03-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Transcatheter Aortic Valve Replacement (TAVR)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prehabilitation Visit/Increased Physical Therapy post-TAVR (Experimental)
  Interventions: Procedure: Prehabilitation visit/increased physical therapy post-TAVR
- Control (Active Comparator): Standard of care physical therapy post-TAVR
  Interventions: Procedure: Standard of Care Arm

INTERVENTIONS:
Procedure: Prehabilitation visit/increased physical therapy post-TAVR — Prior to TAVR, patients randomized to the intervention arm will meet with a licensed physical therapist for a 30-minute session in the ambulatory setting. Following TAVR, patients randomized to the intervention arm will receive 4 days per week of home-based physical therapy by a licensed physical therapist working for Revival Home Health Care
  Arms: Prehabilitation Visit/Increased Physical Therapy post-TAVR
Procedure: Standard of Care Arm — Patients randomized to the usual care arm will receive home-based physical therapy for 2 days per week by Revival Home Health Care, which is the current standard of care.
  Arms: Control

SUMMARY:
The primary purpose of this this randomized interventional study is to determine if increased level of home-based rehabilitation coupled with a pre-TAVR consultation visit in transcatheter aortic valve replacement patients will improve functional status and quality of life and will decrease hospital readmission.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe aortic stenosis (AS) as determined by echocardiography, who are deemed eligible for TAVR by the NYULMC Heart Valve Team

Exclusion Criteria:

* Decisional impairment as assessed by the University of California, San Diego Brief Assessment of Capacity to Consent (UBACC)
* Non-English/non-Spanish speaking.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in level of Activity measured by activity monitor called the ActiGraph wGT3X-BT. | Baseline, 2 Weeks
Change in self-perceived physical health | Baseline, 2 Weeks
Change in Independence in activities of daily living (ADLs). | Baseline, 2 Weeks

SECONDARY OUTCOMES:
Reduction in hospital readmissions following intensive home-based physical therapy reduces | Baseline, 2 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Dodson, MD, Principal Investigator — New York University Medical School